CLINICAL TRIAL: NCT06976281
Title: Effect of Intradialytic Blood Flow Restriction Training on Functional Capacity, Estimated Glomerular Filtration Rate and Health Related Quality of Life in Patients on Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Alaa Sayed Abd El Aziz, principal investigator, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Alaa-02012024
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Blood Flow Restriction Training; Glomerular Filtration Rate; Quality of Life; Hemodialysis
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- blood flow restriction (Experimental): Included 15 chronic kidney disease patients on hemodialysis received conventional exercise program included isometric, aerobic, and resisted exercise individualized for every patient with blood flow restriction by 50% of limb occlusion Pressure. training was conducted for 2 time/weak for 2 consecutive month
  Interventions: Other: conventional exercise Program; Other: blood flow restriction training
- conventional exercise Program (Active Comparator): Included 15 chronic kidney disease patients on hemodialysis received conventional exercise program only included isometric, aerobic, and resisted exercise individualized for every patient. training was conducted for 2 time/weak for 2 consecutive month
  Interventions: Other: conventional exercise Program

INTERVENTIONS:
Other: conventional exercise Program — Exercises include shoulder flexion, shoulder abduction, leg extension, and hand grip. Start with 1-3 sets of 12 reps at 30% of 1-repetition maximum, increasing by 10% according to patient endurance. Cycling is a 30-minute chair or bedside cycle ergometer exercise 2 time/weak for 2 consecutive months
Other: blood flow restriction training — Patients received the same conventional exercise program, which included isometric, aerobic, and resisted exercise individualized for every patient with blood flow restriction by 50% of limb occlusion pressure. Training will be conducted for 2 time/weak for 2 consecutive month
  Arms: blood flow restriction

SUMMARY:
this study was done to investigate the effect of intradialytic blood flow restriction training on functional capacity, estimated glomerular filtration rate and health related Quality of life in patients on Hemodialysis

DETAILED DESCRIPTION:
Chronic kidney disease affects 10% to 15% of the population and is characterized by a progressive decline in glomerular filtration rate. The disease can lead to frailty, muscle mass wasting, and sarcopenia, affecting functional mobility and quality-of-life measures. The increased protein catabolism in Chronic kidney disease is partly due to inflammatory status, nutrient loss during dialysis, and musculoskeletal system changes. Assessment of muscle functionality can provide additional diagnostic and prognostic information for clinical outcomes, quality of life, and mortality rates. Exercise training with blood flow restriction is a potential method for clinical musculoskeletal rehabilitation, potentially improving strength, physical function, blood pressure control, glucose homeostasis, autonomic function, renal deterioration, dialysis adequacy, and antioxidant defenses.

ELIGIBILITY:
Inclusion Criteria:

All patients were

1. Both sex aged from forty to sixty years
2. Stable chronic hemodialysis patient (< 3 months)
3. Participants will be deemed medically eligible by their treating physician before participation in the present study
4. Free from any other disease could interfere with exercise

Exclusion Criteria:

1. Hemodynamic instability during hemodialysis over the last month
2. Neurodegenerative diseases
3. Autoimmune diseases (i.e., lupus erythematosus)
4. Surgery within the past 3 months
5. Severe arrhythmia, angina or cerebrovascular disease
6. Unstable on dialysis
7. Any musculoskeletal problem interfere with exercise

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
assessment of change of estimated glomerular filtration rate | at baseline and after 8 weeks
  Estimated glomerular filtration rate (eGFR) was calculated using the Chronic Kidney Disease Epidemiology Collaboration Creatinine Equation (2021) as recommended by the National Kidney Foundation to assess renal function and detect deterioration.

SECONDARY OUTCOMES:
assessment of change of Limb Occlusion Pressure | at baseline and after 8 weeks
  Limb occlusion pressure was measured using a vascular Doppler ultrasound in combination with a blood flow restriction device to determine individualized occlusion thresholds.
assessment of change of Glucose Homeostasis | at baseline and after 8 weeks
  Glucose regulation was assessed through glycated hemoglobin (HbA1c) levels, reflecting average blood glucose over the previous 2-3 months
assessment of change of upper limb Muscle Strength | at baseline and after 8 weeks
  Upper limb strength was measured using a handgrip dynamometer.
assessment of change of lower limb Muscle Strength | at baseline and after 8 weeks
  lower limb strength was assessed using the One-Repetition Maximum (1RM) test to determine maximum voluntary strength

CONTACTS AND LOCATIONS:
Locations (1):
- out-patient clinic, faculty of physical therapy, beni-suef University, Banī Suwayf, Egypt